CLINICAL TRIAL: NCT00003444
Title: A Prospective Randomized Phase III Clinical Trial Assessing the Role of Post-Operative Radiotherapy Plus Adjuvant Interferon Alpha-2b in Patients With Cervical, Axillary, and Inguinal Nodal Metastasis From Cutaneous Melanoma
Brief Title: Interferon Alfa-2b With or Without Radiation Therapy in Treating Patients With Melanoma That Has Metastasized to Lymph Nodes in the Neck, Under the Arm, or in the Groin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066472; E-3697
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: recombinant interferon alfa
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Interferon alfa-2b may interfere with the growth of cancer cells. It is not yet known whether giving radiation therapy with interferon alfa-2b is more effective than giving interferon alfa-2b alone in treating melanoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy plus interferon alfa-2b with that of interferon alfa-2b alone in treating patients who have melanoma that has metastasized to lymph nodes in the neck, under the arm, or in the groin.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the effectiveness of postoperative hypofractionated radiotherapy in combination with high dose interferon in preventing regional relapse in patients with malignant melanoma with any number of nodes with clinical extracapsular extension or previous nodal basin recurrence. II. Evaluate the effectiveness of this therapy in prolonging relapse free and overall survival in this patient population. III. Evaluate the toxicity of this therapy in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to prior nodal basin recurrence, site of disease, and extracapsular extension. Following surgery, patients are randomized to receive either interferon alfa-2b alone or five treatments of radiotherapy followed by interferon alfa-2b. Patients receive radiotherapy 2 days a week for 2.5 weeks. Patients receive interferon alfa-2b IV over 20 minutes daily for 5 days for a total of 28 days, followed by subcutaneous injections 3 times a week for 48 weeks. Patients are followed every 3 months for 2 years, then every 6 months for 3 years, then annually thereafter.

PROJECTED ACCRUAL: Approximately 167 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented malignant melanoma in node(s) meeting one or more of the following criteria: 1 or more lymph nodes found to contain metastatic melanoma with gross evidence of extracapsular nodal extension Nodal recurrence at the site of previous lymphadenectomy All gross cancer removed with negative margins Prior node biopsy allowed if complete nodal dissection performed Parotid involvement outside a node allowed No distant metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 125,000/mm3 Hematocrit at least 33% Hepatic: AST no greater than 2 times upper limit of normal (ULN) LDH no greater than 2 times ULN Alkaline phosphatase no greater than 2 times ULN Bilirubin no greater than 2 times ULN If LDH or alkaline phosphatase are above normal, CT or MRI of liver required Renal: Creatinine no greater than 1.8 mg/dL BUN no greater than 33 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No other prior or concurrent malignancies within 2 years, except any carcinoma in situ, lobular carcinoma of the breast in situ, carcinoma in situ of the cervix, atypical melanocytic hyperplasia or Clark I melanoma in situ, or basal or squamous cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior interferon Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the head and neck, axillary, or inguinal areas Surgery: See Disease Characteristics Recovered from prior surgery

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 1999-03-29 (Actual); Primary Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maury M. Rosenstein, MD, Study Chair — UPMC Cancer Center at UPMC St. Margaret
Locations (23):
- United States (23):
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin